CLINICAL TRIAL: NCT06718790
Title: The Effect of Menstrual Cup Use on Menstrual Life and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeliha Elkan Kiyat, Research Assistant, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TU-HEM-ZEK-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-12

CONDITIONS: Menstrual Cup
Keywords: Menstrual Cup; Sleep Quality; Menstruation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, there are two groups: menstrual cup users and menstrual pad users
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menstrual cup users (Active Comparator): Women who will use menstrual cups will be trained on the use of the product and a menstrual cup will be provided for them to use. In the next stage, participants will be called by phone in the 1st, 2nd, 3rd and 6th menstrual cycles and asked to answer questions about their menstrual cup use by sharing an online form.
  Interventions: Other: Using menstrual cup
- Menstrual pad users (Active Comparator): For women in the group who will use menstrual pads, the average number of pads they have used in their previous menstrual cycles will be asked and an appropriate number of menstrual pads will be provided. In the next stage, participants will be called by phone in the 1st, 2nd, 3rd and 6th menstrual cycles and asked to answer questions about their menstrual pad use by sharing an online form.
  Interventions: Other: Using menstrual pads

INTERVENTIONS:
Other: Using menstrual cup — In the prospective, randomized controlled study, two groups (Case = Menstrual cup, Control = Menstrual pad) will be randomly formed from individuals who volunteer to participate in the study and meet the inclusion criteria. All participants will be asked to answer the questions in the first interview questionnaire.
  Women who will use menstrual cups will be trained on the use of the product and a menstrual cup will be provided for them to use. In the next stage, participants will be called by phone in the 1st, 2nd, 3rd and 6th menstrual cycles and asked to answer questions about their menstrual cup use by sharing an online form.
  Arms: Menstrual cup users
Other: Using menstrual pads — In the prospective, randomized controlled study, two groups (Case = Menstrual cup, Control = Menstrual pad) will be randomly formed from individuals who volunteer to participate in the study and meet the inclusion criteria. All participants will be asked to answer the questions in the first interview questionnaire. For women in the group who will use menstrual pads, the average number of pads they have used in their previous menstrual cycles will be asked and an appropriate number of menstrual pads will be provided. In the next stage, participants will be called by phone in the 1st, 2nd, 3rd, and 6th menstrual cycles and asked to answer questions about their menstrual pad use by sharing an online form.
  Arms: Menstrual pad users

SUMMARY:
Women's reproductive age is an important process that begins with menarche and ends with menopause. During this period, women need to use safe, effective and affordable products during their menstrual periods. While disposable pads and tampons are the most preferred products today, environmentally friendly and economical options also include menstrual cups, menstrual underwear and reusable pads. Menstrual cups are made of non-toxic silicone or latex, are inserted into the vagina and collect menstrual blood. Studies show that menstrual cups do not have a negative effect on the vaginal flora and most users are satisfied with the product. The environmental impact of menstrual hygiene products should also be taken into account. While disposable pads and tampons harm the environment due to their plastic content, menstrual cups are more sustainable and economical in the long term. In addition, women may experience problems with sleep quality, mood and physical comfort due to the effects of hormones during the menstrual period. However, there is no randomized controlled study yet examining the effects of menstrual cup use on sleep quality and quality of life. The aim of this study was to evaluate the effects of menstrual cup use on menstrual life and sleep quality.

DETAILED DESCRIPTION:
The reproductive age, which constitutes an important part of women's lives, is a process that begins with menarche and continues until menopause. Menstruation is the vaginal discharge of menstrual blood and endometrial tissue during the reproductive age. For women of reproductive age, the menstrual cycle lasts 2-7 days once every 21-35 days on average. Menstrual cycles are generally anovulatory and irregular for at least 2 years following menarche. However, women need to use safe, effective and affordable menstrual products during their menstrual periods. Today, there are many menstrual hygiene products offered to women. Disposable menstrual pads and tampons are the most frequently preferred products. However, new generation products include menstrual cups, menstrual panties, reusable/washable pads and sea sponges. Each of these products has advantages and disadvantages. Menstrual cups, menstrual panties, reusable/washable pads are environmentally friendly and economical products as they can be used for a long time. In addition, pads and tampons are single-use products. While products such as tampons, menstrual cups and sea sponges are placed inside the vagina, pads and menstrual panties are used outside the vagina. However, improper use of menstrual hygiene products can result in health problems such as toxic shock syndrome and risk of infection. Therefore, it is important to have correct information about how to use them.

A woman uses approximately 6000 menstrual pads during her reproductive years. Non-biodegradable waste management consisting of traditional single-use menstrual pads is an important issue for environmental health. In low-income countries, incorrect practices in the disposal of menstrual products cause blockages in sewage pipes and negatively affect sanitation systems. Therefore, menstruation management should also be considered as a public health issue.

Among single-use menstrual hygiene products, single-use menstrual pads in particular affect the environment with their plastic content. In addition, harmful substances such as cyanide, dioxin and bleaches that can negatively affect not only environmental health but also genital health are encountered. In this respect, one of the sustainable menstrual hygiene products that can have less impact on both the environment and genital health is the menstrual cup. A menstrual cup is a reusable menstrual hygiene product that is placed inside the vagina and collects the blood flowing during menstruation. Menstrual cups are usually made of antitoxic silicone or latex. They are also designed in the form of a flexible bell or cup to facilitate women's self-use. There are thoughts that using a menstrual cup may cause toxicity and infection. However, a systematic review and meta-analysis study did not find a negative effect of menstrual cup use on the vaginal flora. However, 5 of the participants reported vaginal pain or sores, 6 allergies or redness, 9 urinary tract complaints and 5 toxic shock syndrome. In the same study, it was reported that 73% of the women using a menstrual cup wanted to continue using the product after the study ended. Sica et al. A study was conducted to evaluate the safety of menstrual cups made of medical silicone. In the study, menstrual cups were evaluated in terms of biocompatibility and chemical safety, physical effect on the vaginal mucosa, effect on the vaginal microbiota and the risk of Staphylococcus aureus growth and toxic shock syndrome. At the end of the study, it was reported that the menstrual cup did not pose a safety problem and was well tolerated. In a study conducted in Kenya, no difference was found in Staphylococcus aureus prevalence in menstrual cup users. One of the factors affecting the use of menstrual hygiene products is economic reasons. Although menstrual cups are expensive when first purchased compared to disposable products, they provide advantages in terms of both cost and solid waste within approximately 6 months of use. During the menstrual period, women may experience problems with mood, body temperature, respiration, autonomic nervous system and sleep regulation due to the effects of reproductive hormones. Sleep problems usually increase in the few days before menstruation and in the first days of menstruation. The cause of sleep problems during the menstrual period may be menstrual period symptoms, menstrual cycle characteristics, or individual-specific reasons. There are limited studies evaluating the menstrual life and sleep quality of women during the menstrual period. Studies conducted focus more on the effects of menstrual symptoms on quality of life. No randomized controlled study has been found examining the effects of menstrual cup use on quality of life and sleep. This study aimed to examine the effects of menstrual cup use on menstrual life and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45,
* Having a regular menstrual cycle between 21-35 days,
* Not having a sexually transmitted disease that has been diagnosed and treated,
* Not having a silicone allergy,
* Not using an intrauterine device,
* Not having a vaginal anatomical defect,
* Not having given birth vaginally (since a standard size menstrual cup will be used)

Exclusion Criteria:

* Those planning to get pregnant,
* Those with a history of sexually transmitted diseases in the last 6 months,
* Those with dysmenorrhea problems will not be included.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | The scale will be used at the end of Cycle 1, 2, 3 and 6 (each cycle is 28 days)
  It was developed to evaluate sleep quality.

SECONDARY OUTCOMES:
Menstruation Impact Scale | The scale will be used at the end of Cycle 1, 2, 3 and 6 (each cycle is 28 days)
  The scale is used to measure the effects of menstruation. Menstruation Impact Scale is a 14-item scale consisting of physical and psychosocial impact subscales. The scale is a 5 point Likert type scale evaluated between "5" Strongly Agree and "1" Strongly Disagree. The minimum and maximum scores to be obtained from the overall scale are 14 and 70 respectively. As the score increases, the participant's degree of being affected by menstruation increases as well.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Elkan Kiyat, Principal Investigator — PhD student
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will be shared upon contact with researchers conducting meta-analysis or systematic reviews.